CLINICAL TRIAL: NCT05979792
Title: Clinical Study of CD7 CAR-T Cell Injection in the Treatment of Patients With Relapsed or Refractory CD7-positive Peripheral T Cell Lymphoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhao Weili (Other)
Responsible Party: Sponsor-Investigator, Zhao Weili, Principal Investigator, Clinical Professor, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHCT-RD13-02P
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T Therapy (Experimental)
  Interventions: Drug: CAR-T Therapy

INTERVENTIONS:
Drug: CAR-T Therapy — CAR-T cell infusion

SUMMARY:
Despite the use of monoclonal antibodies, checkpoint inhibitors, and bispecific T cell adapters (BiTE) Immunotherapies such as chimeric antigen receptor (CAR) T cells have completely changed the treatment methods of various cancers.

However, only limited responses were observed in T cell diseases, In CD30 positive PTCL and CTCL patients. The use of BV in and pembroluzimab (Programmed cell death receptor 1) in the treatment of ENKTL.

Although some promising results have been observed for (PD-1) inhibitors, these positive results are limited to specific subtypes of T cell diseases.

CAR T Cell therapy in recurrent/refractory B-cell malignant tumors is very successful, the Food and Drug Administration (FDA) has approved two CAR T Cell therapy for the treatment of this type of disease. However, using this technology to treat T-cell malignancies has always been difficult, mainly due to the lack of tumor specific surface antigens in cancerous T cells.

Therefore, our center plans to conduct a phase I clinical study of CAR-T to explore the possibility of bringing more treatment options and benefits to PTCL patients.

DETAILED DESCRIPTION:
Patients with recurrent/refractory PTCL were included using a single arm, open label, and single center approach.

Pre treatment plan:

Cyclophosphamide (CTX): 500mg/m2 × 3 days

Fludarabine: 30mg/m2 × 3 days

Note: Researchers can adjust the pre-treatment plan appropriately based on the patient's condition, such as CTX 300mg × Wait for 3 days.

CTX and Flu were infused on the 5th to 3rd day (D-5 to D-3) before administration. RD13-02 can only be injected after 48 hours of pre-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old and<80 years old.
2. According to the clinical practice guidelines for T-cell lymphoma of the National Comprehensive Cancer Network (NCCN) (2022. v2), diagnosis of peripheral T-cell lymphoma, including but not limited to: peripheral T Cell lymphoma, non-specific type (PTCL-NOS), anaplastic large cell lymphoma (ALCL), T helper cell lymphoma (FTCL), peripheral lymph nodes with follicular helper T cell phenotype T-cell lymphoma (TFH) and angioimmunoblastic T-cell lymphoma (AITL), Etc;
3. Relapse or refractory peripheral T-cell lymphoma, which requires at least 2 systematic Sex therapy, is invalid or relapses.
4. Histologically confirmed as CD7 positive.
5. According to Lugano2014 standard, enhanced CT before enrollment should indicate at least one evaluable tumor lesion (with the longest diameter of the intranodal lesion>1.5cm and the longest diameter of the extranodal lesion>1.0cm), and PET/CT should show metabolic activity.
6. Blood routine neutrophil count ≥ 1.0 during screening × 109/L; For individuals without bone marrow invasion, platelet count ≥ 75 × 109/L, Hb ≥ 80g/L; For individuals with bone marrow invasion, platelet count ≥ 50 × 109/L, Hb ≥ 60g/L (if the patient does not meet the screening requirements but meets the screening period requirements for re examination, they can be selected).
7. The average fluorescence intensity (MFI) of donor specific antibodies (DSA) at HLA sites of HLA antibody negative or anti RD13-02 cell derived donors is less than 2000.
8. Creatinine clearance rate>60ml/min (Cockcroft and Gault formula); For patients without liver invasion, serum total bilirubin ≤ 1.5 times the upper limit of normal value, and serum ALT and AST ≤ 3 times the upper limit of normal value range; For patients with liver invasion, serum total bilirubin ≤ 3 times the upper limit of normal value, and serum ALT and AST ≤ 5 times the upper limit of normal value range.
9. Echocardiography showed that left ventricular Ejection fraction (LVEF) ≥ 50%.
10. Estimated survival time of over 3 months.
11. ECOG: 0-1.
12. Subjects or their Legal guardian voluntarily participate in the trial and sign the informed consent form.
13. For patients undergoing reinfusion, in addition to meeting the relevant conditions for reinfusion in the Design of experiments, it is required that there is no DLT event or dose reduction after the first infusion.
14. The first 6 subjects included at any dose level should be able to collect sufficient amounts of autologous hematopoietic stem cells for cryopreservation in advance; Subsequent subjects will be determined by the researcher whether to collect autologous hematopoietic stem cells for cryopreservation.

Exclusion Criteria:

1. Primary cutaneous T-cell lymphoma, including mycosis fungoides (MF) and Sezary syndrome (SS); Enteropathy associated T-cell lymphoma (EATL), monotypic epitheliophagocytic intestinal T-cell lymphoma (MEITL), hepatosplenic T-cell lymphoma (HSTCL), extranodal NK/T-cell lymphoma, nasal type (EENKTCL) and primary central nervous system lymphoma and other types of T-cell leukemia/lymphoma.
2. Active central nervous system (CNS) invasion.
3. If anti-tumor treatment has been received before infusion, it should be excluded if any of the following conditions are met:

   * received small molecule Targeted therapy within 72 hours
   * Received systemic chemotherapy within 2 weeks (excluding pre-treatment)
   * Received radiation therapy within 4 weeks
   * When the time between the last monoclonal antibody infusion and those who have received monoclonal antibody treatment is less than 5 half-lives four weeks long or less (whichever is shorter)
4. Individuals with a history of allergies to any component in cellular products.
5. According to the New York Heart Association (NYHA) cardiac function grading standards, subjects with cardiac dysfunction classified as Class III or IV.
6. Myocardial infarction, cardiac angioplasty or stenting, unstable angina pectoris, or other serious heart disease clinically within 12 months of enrollment.
7. The electrocardiogram indicates that the QT interval is significantly prolonged, and the patient has serious heart disease such as serious arrhythmia in the past.
8. Previous history of craniocerebral trauma, Disorders of consciousness, epilepsy, cerebrovascular ischemia, cerebrovascular hemorrhagic disease, etc.
9. Uncontrolled severe active infections (excluding simple urinary tract infections and bacterial pharyngitis).
10. The subject has a history of other primary cancers, except for the following:

    1. Non Melanoma cured by excision, such as skin Basal-cell carcinoma;
    2. Carcinoma in situ of cervix, local prostate cancer, and ductal Carcinoma in situ with disease-free survival ≥ 2 years after adequate treatment;
11. Subjects with autoimmune diseases requiring treatment or subjects requiring Immunosuppressive drug treatment;
12. Individuals with graft versus host disease (GvHD) and/or requiring immunosuppressive therapy.
13. Live vaccination within 4 weeks prior to screening.
14. The subject has a history of alcoholism, drug abuse, or mental illness.
15. Individuals with EBV DNA copy numbers greater than the upper limit of normal or positive for EBER; CMV copies greater than the upper limit of normal values; HBV or HCV DNA copy number>the upper limit of normal value, and active syphilis or AIDS and other virus infected persons.
16. Subjects who were receiving systemic Sex hormone treatment before screening and who were judged by the investigator to need long-term use of systemic Sex hormone during treatment (except for inhalation or local use).
17. Individuals who have participated in other clinical trials within the first 4 weeks of screening.
18. Pregnant and lactating women and subjects with Fertility who cannot take effective contraceptive measures (both men and women).
19. Any situation that the researcher believes may increase the risk of the subject or interfere with the test results.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Up to 2 years
  DLT

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - The First Affiliated Hospital of USTC, Hefei, Anhui
  - The First Affliliated Hospital of Xiamen University, Xiamen, Fujian
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Affliliated Hospital of Northwest University, Xi’an, Shanxi
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - The 920th Hospital of the Joint Service Support Force of the People's Liberation Army, Kunming, Yunan
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No